CLINICAL TRIAL: NCT01408836
Title: Randomised Trial of Plasma Exchange or High Dose Methyl Prednisolone as Adjunctive Therapy for Severe Renal Vasculitis
Brief Title: Plasma Exchange for Renal Vasculitis
Acronym: MEPEX
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Completed
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University Hospital Birmingham (Other); Imperial College London (Other); London North West Healthcare NHS Trust (Other); University Hospitals, Leicester (Other); Lund University Hospital (Other); University Medical Center Groningen (Other); Fundacio Clinic Barcelona (Other); University of Helsinki (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMH4-CT97-2328
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-07

CONDITIONS: Wegener's Granulomatosis; Microscopic Polyangiitis
Keywords: Vasculitis; ANCA; Therapy; Plasma exchange; Immunosuppression
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Vasculitis | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Plasma exchange x 7 over 14 days
  Interventions: Procedure: Plasma exchange
- 2 (Active Comparator): Methyl prednisolone 1g x 3
  Interventions: Drug: Intravenous methyl prednisolone; Drug: Methyl prednisolone

INTERVENTIONS:
Procedure: Plasma exchange — Plasma exchange
  Arms: 1
Drug: Intravenous methyl prednisolone — Intravenous methyl prednisolone
  Arms: 2
Drug: Methyl prednisolone — methyl prednisolone
  Arms: 2

SUMMARY:
The purpose of this study is to test whether additional therapy with plasma exchange improves the chances of kidney recovery in severe kidney vasculitis.

DETAILED DESCRIPTION:
Primary systemic vasculitis associated with autoantibodies to neutrophil cytoplasmic antigens (ANCA), is the most frequent cause of rapidly progressive glomerulonephritis. Renal failure at presentation often progresses to end stage renal disease despite immunosuppressive therapy. We investigated whether the addition of plasma exchange was more effective than intravenous (IV) methyl prednisolone in the achievement of renal recovery for ANCA associated systemic vasculitis presenting with a serum creatinine above 500umol/l (5.8mg/dl).

137 patients with a new diagnosis of ANCA associated systemic vasculitis, serum creatinine above 500umol/l (5.8mg/dl) and a renal biopsy demonstrating a focal, necrotizing glomerulonephritis were randomized to receive seven plasma exchanges or IV methyl prednisolone 1000mg/day for three days. Both groups were treated with cyclophosphamide and oral prednisolone. The primary end-point was dialysis independence with a serum creatinine below 500umol/l (5.8mg/dl) at three months. Secondary end-points included renal and patient survival at 12 months and severe adverse event rates.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Wegener's granulomatosis or microscopic polyangiitis, using criteria adapted by EUVAS from the disease definitions of the Chapel Hill consensus conference
* Biopsy proven, pauci-immune, necrotising and/or crescentic glomerulonephritis, in the absence of other defined glomerulopathy
* Severe renal impairment defined by: (i) oliguria (<400ml/24hr), or (ii) intention to commence dialysis within 48 hours of admission, and (iii) creatinine >500umol/l (5.8mg/dl).

Exclusion Criteria:

* Age under 18 or over 80 years
* Inadequate contraception in women of child-bearing age
* Pregnancy
* Previous malignancy
* Hepatitis B antigenaemia, anti-hepatitis C virus or anti-human immunodeficiency virus antibody
* Diagnosis of Churg-Strauss syndrome, Henoch-Schönlein purpura, rheumatoid vasculitis, mixed essential cryoglobulinaemia or systemic lupus erythematosus
* Circulating anti-GBM antibodies or linear IgG staining of the GBM on renal biopsy
* Life-threatening non-renal manifestations of vasculitis, including alveolar hemorrhage requiring mechanical ventilation within 24 hours of admission
* On dialysis for > two weeks prior to entry
* Creatinine > 200umol/l (2.3mg/dl) one year or more before entry
* A second clearly defined cause of renal failure
* Previous episode of biopsy-proven necrotising and/or crescentic glomerulonephritis
* > two weeks treatment with cyclophosphamide or azathioprine
* > 500mg IV methyl prednisolone
* Plasma exchange within the preceding year
* > three months treatment with oral prednisolone
* Allergy to study medications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 1995-03; Primary Completion 2003-06 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Renal recovery | Three months

SECONDARY OUTCOMES:
End stage renal disease at 12 months | 12 months
Serum creatinine at 12 months | 12 months
Severe adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Niels Rasmussen, MD, Study Director — Righospitalet, Copenhagen, Denmark
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridge, United Kingdom

REFERENCES:
- [Derived] Walsh M, Casian A, Flossmann O, Westman K, Hoglund P, Pusey C, Jayne DR; European Vasculitis Study Group (EUVAS). Long-term follow-up of patients with severe ANCA-associated vasculitis comparing plasma exchange to intravenous methylprednisolone treatment is unclear. Kidney Int. 2013 Aug;84(2):397-402. doi: 10.1038/ki.2013.131. Epub 2013 Apr 24. PMID 23615499
- See also: EUVAS homepage — http://www.vasculitis.org